CLINICAL TRIAL: NCT00185159
Title: Randomized Olmesartan and Diabetes Microalbuminuria Prevention Study (ROADMAP)
Brief Title: Olmesartan Medoxomil in Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Responsible Party: Heiko Rauer, Daiichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SE-866/44
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Disease; Kidney Disease
Keywords: Microalbuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Kidney Diseases | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): olmesartan medoxomil
  Interventions: Drug: Olmesartan medoxomil
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Olmesartan medoxomil — tablets
  Arms: 1
Drug: Placebo Tablets — Tablets
  Arms: 2

SUMMARY:
This is a study in diabetic patients with at least one additional cardiovascular risk factor and normoalbuminuria prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2, defined as fasting blood glucose of greater than or equal to 126 mg/dL;
* Presence of at least one of the following cardiovascular risk factors:

  1. total cholesterol greater than 200 mg/dL or statin treatment,
  2. High density lipoprotein (HDL) less than 40 mg/dL,
  3. triglycerides greater than 150 mg/dL and less than 400 mg/dL,
  4. blood pressure greater than or equal to 130/80 mmHg,
  5. Body mass index (BMI) greater than 28 kg/m2,
  6. waist circumference greater than 102 cm for men and greater than 88 cm for women,
  7. smoking of more than 5 cigarettes a day;
* Normoalbuminuria at screening

Exclusion Criteria:

* Severe uncontrolled hyperlipidemia;
* Documented renal and/or renal-vascular disease;
* Myocardial infarction, stroke or myocardial revascularization within the last 6 months;
* History of alcohol and/or drug abuse;
* Allergic reaction, lack of response or contraindication to angiotensin receptor blockers (ARBs);
* Current treatment with an ARB or angiotensin converting enzyme (ACE) inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4449 (Actual)
Dates: Start 2004-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Time to the first occurrence of microalbuminuria defined as excretion of greater than 35 mg albumin/g urine creatinine for women and greater than 25 mg albumin/g urine creatinine for men in morning spot urine | Time to the first occurrence

SECONDARY OUTCOMES:
Incidence of cardiovascular mortality and morbidity | Time to occurence
Incidence of renal disease, such as worsening of renal function as well as end-stage (dialysis) | Time to occurrence
Occurrence and progression of retinopathy | Time to occurence
Treatment effects on a combined endpoint of cardiovascular mortality and morbidity and renal disease | Time to occurrence
Safety and tolerability | Throughout entire study

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Hermann Haller, MD, Principal Investigator — Medizinische Hochschule Hannover Klinik fur Nieren, Hannover Germany
Locations (1):
- Darmstadt, Germany

REFERENCES:
- [Derived] Do DV, Han G, Abariga SA, Sleilati G, Vedula SS, Hawkins BS. Blood pressure control for diabetic retinopathy. Cochrane Database Syst Rev. 2023 Mar 28;3(3):CD006127. doi: 10.1002/14651858.CD006127.pub3. PMID 36975019
- [Derived] Chatzikyrkou C, Menne J, Izzo J, Viberti G, Rabelink T, Ruilope LM, Rump C, Mertens PR, Haller H. Predictors for the development of microalbuminuria and interaction with renal function. J Hypertens. 2017 Dec;35(12):2501-2509. doi: 10.1097/HJH.0000000000001491. PMID 29035939
- [Derived] Menne J, Ritz E, Ruilope LM, Chatzikyrkou C, Viberti G, Haller H. The Randomized Olmesartan and Diabetes Microalbuminuria Prevention (ROADMAP) observational follow-up study: benefits of RAS blockade with olmesartan treatment are sustained after study discontinuation. J Am Heart Assoc. 2014;3(2):e000810. doi: 10.1161/jaha.114.000810. PMID 24772521
- [Derived] Menne J, Izzo JL Jr, Ito S, Januszewicz A, Katayama S, Chatzykirkou C, Mimran A, Rabelink TJ, Ritz E, Ruilope LM, Rump LC, Viberti G, Haller H; ROADMAP investigators. Prevention of microalbuminuria in patients with type 2 diabetes and hypertension. J Hypertens. 2012 Apr;30(4):811-8; discussion 818. doi: 10.1097/HJH.0b013e328351856d. PMID 22418908
- [Derived] Haller H, Ito S, Izzo JL Jr, Januszewicz A, Katayama S, Menne J, Mimran A, Rabelink TJ, Ritz E, Ruilope LM, Rump LC, Viberti G; ROADMAP Trial Investigators. Olmesartan for the delay or prevention of microalbuminuria in type 2 diabetes. N Engl J Med. 2011 Mar 10;364(10):907-17. doi: 10.1056/NEJMoa1007994. PMID 21388309
- [Derived] Januszewicz A, Ritz E, Viberti G, Mimran A, Rabelink AJ, Rump LC, Ruilope LM, Katayama S, Ito S, Izzo JL Jr, Haller H. Office and ambulatory pulse pressure--association with clinical characteristics and cardiovascular risk factors in normoalbuminuric patients with type 2 diabetes (ROADMAP study). J Hum Hypertens. 2011 Nov;25(11):679-85. doi: 10.1038/jhh.2010.111. Epub 2010 Dec 9. PMID 21150933
- [Derived] Ritz E, Viberti GC, Ruilope LM, Rabelink AJ, Izzo JL Jr, Katayama S, Ito S, Mimran A, Menne J, Rump LC, Januszewicz A, Haller H. Determinants of urinary albumin excretion within the normal range in patients with type 2 diabetes: the Randomised Olmesartan and Diabetes Microalbuminuria Prevention (ROADMAP) study. Diabetologia. 2010 Jan;53(1):49-57. doi: 10.1007/s00125-009-1577-3. Epub 2009 Oct 30. PMID 19876613